CLINICAL TRIAL: NCT06184282
Title: Assessment of Topical Mebo Versus Lidocane in Healing Time of Traumatic Oral Ulcer: Randomized Controlled Trial
Brief Title: Topical Mebo Versus Lidocane in Healing Time of Traumatic Oral Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Amany Ahmed Mohamed Alaraby, Lecturer of Oral Medicine, Diagnosis and Periodontology, Faculty of Dentistry, October 6 University, 6 October city, Egypt, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECO6U/15-2023
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Mebo; Lidocaine; Healing; Traumatic Oral Ulceration
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEBO group (Experimental): MEBO (Julphar®, Ras Al Khaimah, United Arab Emirates) was applied using sterile plastic brush daily and the patients were recalled at 2, 5 and 10 days for evaluating the healing of the ulcer.
  Interventions: Drug: MEBO
- Control Group (Active Comparator): Lidocaine gel was applied using sterile plastic brush daily and the patients were recalled at 2, 5 and 10 days for evaluating the healing of the ulcer.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: MEBO — MEBO (Julphar®, Ras Al Khaimah, United Arab Emirates) was applied using sterile plastic brush daily and the patients were recalled at 2, 5 and 10 days for evaluating the healing of the ulcer.
  Arms: MEBO group
Drug: Lidocaine — Lidocaine gel was applied using sterile plastic brush daily and the patients were recalled at 2, 5 and 10 days for evaluating the healing of the ulcer.
  Arms: Control Group

SUMMARY:
This study aims to assess topical MEBO application on pain relief and wound healing.

DETAILED DESCRIPTION:
One of the conditions that affect the mouth frequently is a traumatic ulcer. Between 3 and 24 % of the population are affected, which is a significant prevalence. It is symptomatic to treat traumatized ulcers. Oral wound healing is a dynamic process and complicated phenomenon involving secondary concerns, a succession of overlapping stages of rebuilding cell and tissue structure.

Inflammation, granulation tissue creation, matrix formation, re-epithelialization, and tissue remodeling are some of the cellular and physiological activities that occur during wound healing.

Oral wound healing is a dynamic process and complex phenomenon involving secondary issues, series overlapping stages of restoring tissue and cellular structures.

Since 1995, the Moist Exposed Burn Ointment (MEBO), a Chinese burn ointment, has had a recognized US patent. Beta-sitosterol, Phellodendron amurense, Scutellaria baicalensis, Coptis chinensis, Pheretima aspergillum, Beeswax, and sesame oil are all natural ingredients found in MEBO, a pure herbal extract.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 50 years.
* Both sexes.
* Systemically healthy patients.
* Patients with good oral hygiene.

Exclusion Criteria:

* Patients with any uncontrolled local or systemic disease.
* Smokers.
* Pregnancy and lactation.
* Patients allergic to the used agents.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
The degree of pain | 10 days after surgery
  Pain score was reported by the patient directly through Visual Analogue Scale (VAS) score (between 0 and 10; 0: no pain, 1:minimal pain, 5: moderate pain, and 10: severe pain) VAS was recorded daily for 1 week.

SECONDARY OUTCOMES:
Wound Size | 10 days after surgery
  Wound size was measured using (UNC-15) periodontal probe. Wound size was measured at baseline and on days 2, 5, and 10.
The degree of re-epithelization | 10 days after surgery
  Cytological analysis was performed using the superficial epithelial cell index indices at 2, 5 and 10 days.
  Superficial cell index = Cells with or without pyknotic nuclei / Total no. of examined cells x100
The degree of keratinization | 10 days after surgery
  Cytological analysis was performed using keratinization indices at 2, 5 and 10 days.
  Keratinization index = Cells without nuclei / Total no. of examined cells x100

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.